CLINICAL TRIAL: NCT07238179
Title: Side Effects of a Single Shot Intrathecal Morphine in Clinical Practice, a Retrospective Analysis
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s70568
Record Dates: First submitted 2025-09-24; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Morphine; Morphine Adverse Reaction; Morphine Induced Pruritis; Nausea and Vomiting, Postoperative; Analgesia; Spinal Analgesia
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intrathecal morphine
  Interventions: Drug: Intrathecal Morphine

INTERVENTIONS:
Drug: Intrathecal Morphine — The administration of intrathecal morphine (2µg/kg, with a maximum of 150-200µg) according to standard practice in a variety of surgical procedures. In addition, patients of 2 RCT using 4 or 5µg/kg (max 400 or 500µg), will also be included.

SUMMARY:
ITM has the potential to be a powerful tool for multimodal postoperative pain management, understanding, preventing and managing its side effects is crucial for upturn of patient safety and comfort. This retrospective audit will therefore be focused on the most reported side effects in daily clinical practice in patients having received ITM. The results of this study may lead to new insights into the clinically relevant risk-benefit balance of ITM and will contribute to the optimisation of its use in clinical practice.

DETAILED DESCRIPTION:
Most patients undergoing invasive procedures experience postoperative pain. The definition of pain is described as an unpleasant sensory and emotional experience associated with actual or potential tissue damage or described in terms of such damage. Postoperative incisional pain is a unique and common form of acute pain. Recent studies demonstrate that about 50-70% of patients experience moderate to severe pain after surgery indicating that postoperative pain remains poorly treated.

Mismanagement of acute postoperative pain compromises patient recovery by increasing morbidity and delaying recovery. Therefore, adequate pain treatment is crucial. Steps for formulating a multimodal regimen consider both non pharmacologic and pharmacologic therapies. Opioids are considered a staple in the management of acute postoperative pain. Opioid analgesics embody a wide range of medicinal products that share the ability to relieve acute severe pain by acting on the opioid receptors. There has been a significant increase in the number of opioid analgesics, and they differ in their chemical composition and route of administration (oral, intravenous, subcutaneous, intramuscular, topical, transmucosal, transdermal, neuraxial). Despite their effectiveness in pain relief, opioids are also associated with side effects, including physical dependence and respiratory depression. Consequently, researchers have been exploring alternative methods of opioid administration to minimise the risk of these side effects, one of which is intrathecal opioid delivery.

Since their introduction in the 1970s, intrathecal opioids have been extensively utilised and have gained significant popularity for their efficacy in the management of postoperative pain. Intrathecal morphine (ITM) refers to the single injection of morphine into the subarachnoid space between two lumbar vertebrae. It can be used in combination with general anaesthesia, as adjuncts to intrathecal local anaesthetics or alone. It is rather easy to administer and when used as a single shot technique, it can provide long-lasting effective postoperative analgesia. Moreover, it can decrease systemic opioid consumption and potentially facilitates enhanced recovery due to optimised pain management and faster mobilisation.

Despite its potential, the use of ITM is restrained in daily clinical practice due to the concerns about the potential side effects, including postoperative nausea and vomiting (PONV), pruritus, urinary retention, sedation and respiratory depression. Especially the latter is a reason for clinicians to be reluctant to the use of ITM. At present, data regarding the incidence and severity of side effects following ITM is relatively limited. Respiratory depression is one of the most serious side effects and appears to be dose dependent. Since lower doses of ITM are currently being used, it occurs less frequently than in the past. Respiratory depression has no clear definition in the literature and can be caused by several factors, which makes it challenging to investigate. Studies report an incidence ranging from 0 to 3.4%, depending on the dose of ITM. A single shot up to 150µg seems to be safe and the risk of respiratory depression equals that of systemic opioids in this dosage. A higher amount of ITM may increase the risk of respiratory depression, without necessarily improving analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery and receiving general anaesthesia with preoperative administration of a single shot of ITM.

Exclusion Criteria:

* Patients who are less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient receiving intrathecal morphine and combined with general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of respiratory depression in the first 24 hours postoperatively | 24 hours postoperatively
  Incidence of respiratory depression defined as followed:
  * Prolonged intubation and ventilation (>2 hours) despite adequate reversal of neuromuscular block. OR
  * Support of ventilation following extubation with either non-invasive or invasive ventilation. OR
  * Primary respiratory acidosis (in an extubated patient). OR
  * Reporting of bradypnea, respiratory rate < 8/min.

SECONDARY OUTCOMES:
Number of patients reporting pruritus within the first 24 hours postoperatively | First 24 hours postoperatively
  Based on the electronic health records we will identify whether there is a reporting of patients experiencing pruritus or received treatment for pruritus (administration of antihistamines).
Number of patients reporting clinically relevant postoperative nausea and vomiting within the first 24 hours postoperatively | First 24 hours postoperatively
  Based on the electronic health record, we will identify patients with PONV numeric rating scale (NRS) score >3 (on a scale from 0-10) and/or receiving additional treatment with anti-emetics.
Incidence of patient requiring urinary retention bladder catheterization during their stay on the post-anesthesia care unit or up to 24 hours postoperatively. | First 24 hours postoperatively
  Using the electronic health record we will identify the patients requiring bladder catheterization during their stay on the post-anesthesia care unit or on the normal ward up till 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Danny F Hoogma, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Pseudoanonymised data will be available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Following publication until 3 years later
Access Criteria: Contact the PI